CLINICAL TRIAL: NCT00871858
Title: Response to Neoadjuvant Treatment With Anti-aromatase Anastrozole and Anti-estrogen Fulvestrant: a Randomized Phase II Study in Postmenopausal Patients With Hormone-sensitive Non-metastatic Breast Cancer and an Exploratory Study of Molecular Signatures of Response.
Brief Title: Anastrozole or Fulvestrant in Treating Postmenopausal Patients With Breast Cancer
Acronym: HORGEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633329; 2007-004216-31 (EudraCT Number)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (ANA) (Active Comparator): Patients receive oral anastrozole as 1 mg film-coated tablets, once daily for 6 months.
  Interventions: Drug: anastrozole
- Arm B (FULV) (Experimental): Patients receive fulvestrant intramuscularly ( 250 mg/5 ml solution) on days 1, 14, and 28 and then once a month thereafter until 6 months.
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: anastrozole — Given orally
  Arms: Arm A (ANA)
Drug: fulvestrant — Given intramuscularly
  Arms: Arm B (FULV)

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using anastrozole may fight breast cancer by lowering the amount of estrogen the body makes. Fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. Given the lack of clinical data on fulvestrant in patients with large operable or locally advanced hormone-receptor-positive breast cancer, and the potential to identify differences in the mechanism of resistance using the neoadjuvant model,we decided to perform a multicentre randomised phase II clinical trial of anastrozole and fulvestrant.

PURPOSE: The aim of this study was to assess the efficacy of neoadjuvant anastrozole and fulvestrant treatment of large operable or locally advanced hormone-receptor-positive breast cancer not eligible for initial breast-conserving surgery, and to identify genomic changes occurring after treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate clinical tumor response at 6 months in patients with hormone-sensitive non-metastatic breast cancer treated with neoadjuvant anastrozole and fulvestrant.

Secondary

* Evaluate tumor regression by mammography and ultrasound in these patients.
* Evaluate the rate of breast conservation at 6 months of treatment in these patients.
* Evaluate the tolerability of these regimens.
* Estimate the relapse-free survival at 5 years.
* Identify molecular signatures predictive of response in these patients.
* Identify genes implicated in response in these patients.
* Identify changes in mRNA splicing of genes involved in breast tumorigenesis.

OUTLINE: This is a non-comparative multicentre randomised phase II study in which patients from three French centres were randomly assigned in a 1 : 1 ratio to receive either anatrozole or fulvestrant.

All patients undergo biopsy at baseline. Patients are randomized between the two treatment arms.

* Arm I: Patients receive oral anastrozole once daily for 6 months.
* Arm II: Patients receive fulvestrant intramuscularly on days 1, 14, and 28 and then once a month at 2-6 months.

Within 8 days after completion of hormone therapy, all patients undergo surgical resection of the residual lesion followed by radiotherapy. Patients then receive oral anastrozole once daily for 5 years.

Tissue samples from biopsy and surgery are analyzed to assess molecular signatures and sensitivity to treatment, and to compare gene expression variation with response.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer, meeting 1 of the following criteria:

  * SBR grade I-II disease (patients < 65 years of age)
  * SBR grade I-III disease (patients > 65 years of age)
* T2 (2-5 cm), T3, or T4B, and N0-1 disease
* No metastatic disease
* Breast lesion not amenable to breast-conserving resection
* No inflammatory breast cancer
* No prior breast cancer
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive

PATIENT CHARACTERISTICS:

* Postmenopausal
* No other cancer within the past 5 years except for adequately treated skin carcinoma or carcinoma in situ of the cervix
* No contraindication to anti-hormonal treatment
* No psychological, familial, social, or geographical reasons that would preclude follow up

PRIOR CONCURRENT THERAPY:

* At least 8 days since prior hormone replacement therapy
* No concurrent anti-vitamin K treatment

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03-18 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Mauriac, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

REFERENCES:
- [Result] Quenel-Tueux N, Debled M, Rudewicz J, MacGrogan G, Pulido M, Mauriac L, Dalenc F, Bachelot T, Lortal B, Breton-Callu C, Madranges N, de Lara CT, Fournier M, Bonnefoi H, Soueidan H, Nikolski M, Gros A, Daly C, Wood H, Rabbitts P, Iggo R. Clinical and genomic analysis of a randomised phase II study evaluating anastrozole and fulvestrant in postmenopausal patients treated for large operable or locally advanced hormone-receptor-positive breast cancer. Br J Cancer. 2015 Aug 11;113(4):585-94. doi: 10.1038/bjc.2015.247. Epub 2015 Jul 14. PMID 26171933
- [Derived] Lerebours F, Pulido M, Fourme E, Debled M, Becette V, Bonnefoi H, Rivera S, MacGrogan G, Mouret-Reynier MA, de Lara CT, Pierga JY, Breton-Callu C, Venat-Bouvet L, Mathoulin-Pelissier S, de la Motte Rouge T, Dalenc F, Sigal B, Bachelot T, Lemonnier J, Quenel-Tueux N. Predictive factors of 5-year relapse-free survival in HR+/HER2- breast cancer patients treated with neoadjuvant endocrine therapy: pooled analysis of two phase 2 trials. Br J Cancer. 2020 Mar;122(6):759-765. doi: 10.1038/s41416-020-0733-x. Epub 2020 Jan 31. PMID 32001832

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (ANA) | Arm B (FULV)
Started | 61 | 59
Evaluable for Safety | 60 (1 patient refused to continue study and therefore did not received treatment.) | 58 (1 patient refused to continue study after randomization and therefore did not received treatment.)
Completed | 56 | 52
Not Completed | 5 | 7
Not completed — Protocol Violation | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (ANA) | Arm B (FULV) | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.1 [64.1 to 77.5] | 70.5 [64.0 to 77.8] | 69.8 [64.0 to 77.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 120
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Determined by Clinical Palpation
Description: Objective response rate is defined as the rate of participants with partial or complete responses according to RECIST V1.0.
  Complete response is defined as the disappearance of all target lesions and partial response is defined as at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD (RECIST V1.0.).
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ANA) | Arm B (FULV)
Number analyzed (Participants) | 56 | 52
percentage of participants | 58.9 [45.0 to 71.9] | 53.8 [39.5 to 67.8]

2. Secondary Outcome: Objective Response Rate (ORR) Determined by Ultrasound
Description: as for outcome 1
Time Frame: 6 months
Population: Out of 108 patients (56 arm A + 52 arm B) evaluable for efficacy ("completed" in flow chart) : 19 patients in Arm A and 31 in arm B with missing size at ultrasound examination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ANA) | Arm B (FULV)
Number analyzed (Participants) | 37 | 21
percentage of participants | 35.1 [20.2 to 52.5] | 52.4 [29.8 to 74.3]

3. Secondary Outcome: Objective Response Rate (ORR) Determined by Mammography
Description: as for outcome 1
Time Frame: 6 months
Population: Out of 108 patients (56 arm A + 52 arm B) evaluable for efficacy ("completed" in flow chart) : 33 patients in Arm A and 34 in arm B with missing size at mammography.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ANA) | Arm B (FULV)
Number analyzed (Participants) | 23 | 18
percentage of participants | 26.1 [10.4 to 48.4] | 27.8 [9.7 to 53.5]

4. Secondary Outcome: Rate of Breast-conserving Surgery
Description: breast-conserving surgery concerns patients who did not undergo mastectomy.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ANA) | Arm B (FULV)
Number analyzed (Participants) | 56 | 52
percentage of participants | 60.7 [46.8 to 73.5] | 50.0 [35.8 to 64.2]

5. Secondary Outcome: Percentage of Participants With 5-year Relapse-Free Survival
Description: Relapse-Free survival (RFS) is measured from the date of randomization to the date of the following events, whichever occurs first according to the DATECAN recommendations for breast cancer:
  * Invasive ipsilateral breast tumor recurrence/ progression ;
  * Local invasive recurrence/progression ;
  * Regional invasive recurrence/progression (N+: regional progression) ;
  * Appearance/Occurrence of Metastatic recurrence;
  * Death whatever the cause.
  Participants who did not experience events were censored at the date of last follow-up. RFS was estimated using the Kaplan-Meier method. No comparison test was performed between the two arms as this study is non-comparative.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A (ANA) | Arm B (FULV)
Number analyzed (Participants) | 56 | 52
Percentage of participants | 82.8 [69.6 to 90.7] | 74.7 [60.4 to 84.5]

ADVERSE EVENTS:
Arm/Group | Arm A (ANA) | Arm B (FULV)
All-Cause Mortality (participants affected / at risk) | 6/60 | 6/58
Serious Adverse Events (participants affected / at risk) | 2/60 | 3/58
Other Adverse Events (participants affected / at risk) | 48/60 | 43/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (ANA) (N=60) | Arm B (FULV) (N=58)
Clear cell kidney cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endometrial atrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Programmed peritoneal dialysis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (ANA) (N=60) | Arm B (FULV) (N=58)
Fatigue (General disorders) | 7 (7) | 19 (20) — SOC CTCAE V3.0 = constitutional symptoms
Weight gain (Investigations) | 3 (3) | 2 (2) — SOC CTCAE V3.0= Constitutional symptoms
Injection site reaction (General disorders) | 0 (0) | 9 (9) — SOC CTCAE V3.0= Dermatology/Skin
Hot flashes (Vascular disorders) | 13 (13) | 14 (14) — SOC CTCAE V3.0=Endocrine gastrointestinal
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) — SOC CTCAE V3.0= Neurology
Agitation (Psychiatric disorders) | 3 (3) | 4 (4) — SOC CTCAE V3.0=Neurology / AE term CTCAE V3.0= Mood alteration
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (20) | 11 (11) — SOC CTCAE V3.0=PAIN
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — SOC CTCAE V3.0= PAIN

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes